CLINICAL TRIAL: NCT01708772
Title: The Predictive Prognostic Values of Serum TNF-a in Comparison to SOFA Score Monitoring in Critically Ill Patients
Brief Title: Serum TNF-a in Comparison to Sequential Organ Failure Assessment (SOFA) Score Monitoring in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant Professor of Anesthesia, Tanta University
Other Study IDs: 1381/09/12
Record Dates: First submitted 2012-10-10; First posted 2012-10-17 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Sepsis; Critically Ill
Keywords: TNF alpha; SOFA score
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis: Forty five patients developed septic complication during ICU stay (sepsis group).
- SIRS group: Forty five patients were critically ill without evidence of infectious organism (SIRS group).

SUMMARY:
A total of ninety patients (52men and 38women) were included in the study. Forty five patients developed septic complication during ICU stay (sepsis group). Forty five patients were critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis were measured. Routine cultures were obtained. The attending physician evaluated the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of TNF-a and SOFA score was monitored.

DETAILED DESCRIPTION:
The patients staying in ICU for more than 24 hours were enrolled in the study. Patients received anti-inflammatory drugs or corticosteroids before admission, patients had immunosuppressive illness, patients had chronic organ failure; patients received massive blood transfusion; patients with radiation therapy and patients with previous organ transplantation were excluded from the study. At admission, patient's age, sex, weight and height were recorded. Patients data that include the clinical status; sequential organ failure assessment (SOFA) score; temperature; heart rate; respiratory rate; blood pressure; central venous pressure; laboratory analysis (complete blood count, blood urea nitrogen, blood sugar, serum sodium, potassium, calcium, aspartate aminotransferase, alanine aminotransferase, prothrombin time, albumin and CRP) and arterial blood gas analysis were measured. Routine cultures of suspected sites, blood and urine were obtained to determine the presence of infection. We attempted to maintain the patient hemoglobin level at 10-12g/dl and central venous pressure at 8-12 cmH2o. When needed, intravascular fluid replacement, blood products and inotropic or vasopressor agents were administered. Each day the attending physician evaluated all the study patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU.

ELIGIBILITY:
Inclusion Criteria:

* The patients staying in ICU for more than 24 hours were enrolled in the study.

Exclusion Criteria:

* The Patients received anti-inflammatory drugs or corticosteroids before admission, patients had immunosuppressive illness, patients had chronic organ failure;
* Patients received massive blood transfusion;
* Patients with radiation therapy and patients with previous organ transplantation were excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of ninety patients (52men and 38women) were included in the study. Forty five patients developed septic complication during ICU stay (sepsis group). Forty five patients were critically ill without evidence of infectious organism (SIRS group). Patients were classified into their groups at the time of the first blood analysis for these biomarkers at ICU admission.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
TNF-a determination using ELISA. | Participants will be followed for the duration of ICU stay, At admission, 3rd, 5th and 7th day of ICU stay.Patients will be followed for at least 2 weeks.
  A serum level of TNF-a was determined by quantitative sandwich enzyme immunoassay (R&D Systems, Inc., Minneapolis, MN, USA) guided by to the manufacturer's instructions. The intensity of the color was measured at 490 nm.

SECONDARY OUTCOMES:
Evaluation of SOFA score: | Participants will be followed for the duration of ICU stay, at admission, 3rd, 5th, and 7th day of ICU stay.Patients will be followed for at least 2 weeks.
  SOFA score is composed of scores of six organ systems (respiratory [R], cardiovascular [C], hepatic [H], coagulation [Co], renal [Re], and neurological [N]) graded from 0 to 4 according to the degree of dysfunction/ failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant professor os Anesthesia and ICU, Faculty of Medicine, Tanta university
Locations (1):
- Tanta university, Tanta, Algharbiya, Egypt

REFERENCES:
- [Background] Ferrerira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA 2001:286(14):1754-1758. Sheeran P, Hall GM. Cytokine balance and immunosuppressive changes at cardiac surgery. Br J Anaesth 1996; 77: 129-30. Robertshaw H J, Brennan F M. Release of tumour necrosis factor a (TNF-a) by TNF a cleaving enzyme (TACE) in response to septic stimuli in vitro. Br J Anaesth 2005; 94: 222-8.